CLINICAL TRIAL: NCT01229553
Title: Effect of Topical and Systemic Decolonization of Staphylococcus Aureus (SA) in Pediatric Cystic Fibrosis (CF) Patients at the CF Center at SUNY Upstate Medical University, Syracuse, NY.
Brief Title: Effect of Topical and Systemic Decolonization of Staphylococcus Aureus (SA) in Pediatric Cystic Fibrosis (CF) Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol was never implemented as procedures became standard of care
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Jana Shaw/ MD, MPH, FAAP, Assistant Professor, SUNY Upstate Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5975
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decolonization group (Experimental): The decolonization protocol for the patients will consist of two-week course of cephalexin (100 mg/kg/day divided TID) or oral T/S (20 mg/kg/day divided BID), HBW every other day for 2 weeks, and mupirocin ointment into both nares BID for 2 weeks.
  Interventions: Drug: decolonization

INTERVENTIONS:
Drug: decolonization — The decolonization protocol for the patients will consist of two-week course of cephalexin (100 mg/kg/day divided TID) or oral T/S (20 mg/kg/day divided BID), HBW every other day for 2 weeks, and mupirocin ointment into both nares BID for 2 weeks.

SUMMARY:
The primary objective of this study is to measure efficacy of our new protocol by monitoring the results of our routine respiratory cultures at the end of the new standard treatment, and during routine visits for 1 year from initiation of therapy for Staphylococcus aureus. The secondary objective will include determining the clinical course (pulmonary exacerbations, antibiotic use, hospitalizations, pulmonary function tests) of patients who underwent the protocol.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will include all patients with CF who test positive for SA from respiratory tract culture (throat, nares or expectorated sputum) and are 2-23 months of age at protocol presentation.

Exclusion Criteria:

Patients co-infected with other bacteria (e.g. Pseudomonas) or documented to have an allergy or resistance to any of the intervention substances will be excluded.

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To measure the efficacy of a decolonization regimen to eliminate SA from nares, oropharynx and sputum of pediatric CF patients (2-23 months of age). | 1 year

SECONDARY OUTCOMES:
To measure adverse effects of the decolonization regimen (e.g. local irritation, skin dryness, rashes, vomiting, diarrhea) and its impact on carriage with other organisms (e.g., Pseudomonas). | 1 year
To evaluate the effect of decolonization regimen on lung changes and/or frequency of pulmonary exacerbations. | 1 year
To evaluate adherence to the decolonization regimen | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jana Shaw, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States